CLINICAL TRIAL: NCT06602830
Title: I-gel Plus Supraglottic Airway Device for Elective Laparoscopic Surgery -a Prospective Observational Study-
Brief Title: I-gel Plus Supraglottic Airway Device for Elective Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-101346-BO-ff
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Airway Management; Supraglottic Airway; General Anesthesia; Laparoscopic Surgery
Keywords: Airwaymanagement; Laparoscopic surgery; Capnoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing laparoscopic surgery: Measurement of primary and secondary outcome parameters at different time points during the procedure.

SUMMARY:
i-gel Plus is a novel supraglottic airway device (SGA). Feasibility of second-generation SGAs in patients undergoing elective laparoscopic surgery has been demonstrated in various studies. During laparoscopic surgery intrabdominal pressure is increased by capnoperitoneum and frequently minute ventilation has to be adopted to counteract hypercapnia, and higher inspiratory peak pressures have to be expected. It is uncertain, however, if the i-gel Plus facilitates appropriate ventilation with low leakage volumes in patients undergoing laparoscopic surgery.

The primary aim of this single-center non-inferiority study is to assess the leak fraction of the i-gel Plus under conditions of capnoperitoneum (with and without Trendelenburg position) and to compare it with baseline conditions. Secondary aims are to assess secondary outcome parameters during capnoperitoneum (with and without Trendelenburg position) and to compare them with baseline conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduling for elective laparoscopic surgery
* Planned airway management using a SGA
* Adult patients (age 18-89 years)
* ASA physical status 1-3

Exclusion Criteria:

* Pregnant or breastfeeding women
* Non-fasted patients
* Increased risk of aspiration or other contraindications for supraglottic mask ventilation
* Body mass index (BMI) >35 kg/m2
* Inability to understand or sign informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic surgery with i-gel Plus used for airway management
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Leak fraction | 3 houres
  Ventilation parameter - volume per tidal volume

SECONDARY OUTCOMES:
Oropharyngeal seal pressure [cm H2O] | 3 houres
  Clinical assessment - leak pressure with audible leak
Leakage volume (ml) | 3 houres
  Ventilation parameter - as displayed on the ventilator
Tidal volume (ml) | 3 houres
  Ventilation parameter - as displayed on the ventilator
Inspiratory peak pressure (cm H2O) | 3 houres
  Ventilation parameter - as displayed on the ventilator
Positive endexpiratory pressure (PEEP) (cm H2O) | 3 houres
  Ventilation parameter - as displayed on the ventilator
Intraabdominal pressure under capnoperitoneum [mmHg] | 3 houres
  Measured intraoperativ under capnoperitoneum [mmHg]
Respiratory rate (1/min) | 3 houres
  Ventilation parameter - as displayed on the ventilator
Minute ventilation (l/min/kg) | 3 houres
  Ventilation parameter - as displayed on the ventilator
Endtidal CO2 [mmHg] | 3 houres
  Ventilation parameter - as displayed on the ventilator
Number of insertion attempts | 3 houres
  Clinical assessment - SGA insertion attempts
Insertion success rate (%) | 3 houres
  Clinical assessment
First-attempt insertion success rate (%) | 3 houres
  Clinical assessment - successful placement in only one insertion attempt
Necessity of adjustment maneuvers during the procedure | 3 houres
  Clinical assessment
Insertion time (sec) | 3 houres
  Clinical assessment
Lowest oxygen saturation (%) | 3 houres
  Measured by pulse oximetry
Difficulty of insertion | 3 houres
  Clinical assessment on a scale between 1-5
Ease of gastric tube insertion | 3 houres
  Clinical assessment - rating on a scale from 1-5
Postoperative complications | 24 hours postoperatively
  Clinical assessment
Complications at the end of surgery | 3 hours
  Clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany